CLINICAL TRIAL: NCT06128434
Title: Clinical and Laboratory Effectiveness of Different Toothpastes in Treating White Spot Lesions
Brief Title: Effectiveness of Different Toothpastes in Treating White Spot Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M08040521
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-11

CONDITIONS: White Spot Lesions [Initial Caries] on Smooth Surface of Tooth

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial involving 21 participants ages 12 to 18 years. They will be examined and chosen randomly for the study. Participants will be divided equally into three groups: Group 1 will use zinc carbonate nano-hydroxyapatite toothpaste twice daily; Group 2 will apply 8% arginine and calcium carbonate-containing toothpaste twice daily; and Group 3 will apply fluoridated toothpaste twice daily. Assessment of white spot lesions will be carried out using digital photographs before remineralizing agent application (baseline) and at 3, and 6 month intervals.
Who Masked: Participant, Outcomes Assessor
Masking Description: The toothpastes are sourced from international markets, and both the participants and the outcome assessor will remain unaware of the active remineralizing agent in the toothpaste. This ensures that neither the participants nor the outcome assessor will be informed about the assigned intervention, preventing their expectations from influencing the study results.
  The examiner was blinded to participants' codes and previous WSL scores during dental assessments. However, blinding to the type of toothpaste used was not possible. Blinding during image analysis was also unfeasible, but this limitation was deemed manageable since the outcome relied on objective computer-based data, minimizing potential bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- zinc carbonate nano-hydroxyapatite toothpaste (Experimental): Biorepair toothpaste with 20 wt% zinc carbonate nano-hydroxyapatite
  Interventions: Other: zinc carbonate nano-hydroxyapatite toothpaste
- 8% arginine toothpaste (Experimental): Colgate Sensitive Pro-Relief™ with pro-argin technology
  Interventions: Other: 8% arginine toothpaste
- Fluoride toothpaste (Active Comparator): Signal cavity fighter toothpaste with Sodium Monofluorophosphate
  Interventions: Other: Fluoride toothpaste

INTERVENTIONS:
Other: zinc carbonate nano-hydroxyapatite toothpaste — Participants will brush their teeth with zinc carbonate nano-hydroxyapatite toothpaste twice daily.
  Other Names: Biorepair
  Arms: zinc carbonate nano-hydroxyapatite toothpaste
Other: 8% arginine toothpaste — Participants will brush their teeth with 8% arginine toothpaste twice daily.
  Other Names: Colgate Sensitive Pro-Relief™
  Arms: 8% arginine toothpaste
Other: Fluoride toothpaste — Participants will brush their teeth with Fluoride toothpaste twice daily.
  Other Names: signal cavity fighter
  Arms: Fluoride toothpaste

SUMMARY:
This randomized clinical trial and laboratory study was conducted to:

Compare the effectiveness of zinc-carbonated nano-hydroxyapatite, arginine, and fluoride-containing toothpastes for treating white spot lesions associated with orthodontically treated teeth by using:

* Computerized image software analysis.
* Energy dispersive X-ray analysis.

DETAILED DESCRIPTION:
White spot lesions (WSLs), defined as "white opacity," occur as a result of subsurface enamel demineralization that is located on smooth surfaces of teeth. The reason for the white appearance is the changes in light-scattering optical properties of the decalcified enamel. The aim of the current study is to compare the effectiveness of zinc-carbonated nano-hydroxyapatite, arginine, and fluoride-containing toothpastes for treating white spot lesions.

A) Primary Objective

Assessment of:

size and color change measurements of the WSLs through digital photography and computerized image software analysis.

B) Secondary Objectives

Assessment of:

* Degree of remineralization using Energy dispersive X-ray analysis

PICOTS:

• P - Participants: patients in the age group of 12-18 years having post orthodontic white spot lesions (WSLs).

I - Intervention:

* zinc-carbonated nano-hydroxyapatite-containing toothpaste.
* 8% arginine and calcium carbonate-containing toothpaste (Pro-Argin technology)

C- Comparison:

fluoride-containing toothpaste.

O -Outcomes:

* Reduction in WSLs size and color improvement
* remineralization of WSLs by regaining Ca and P ions.

T- Time: study period will be over 6 months.

S- Study design: Randomized Controlled Trial (RCT) and in vitro study

This study will consist of two parts: in vivo part (Randomized Controlled Trial) and in vitro part:

In vivo part:

* Study design: Randomized controlled trial (RCT)
* Grouping:

Patients will be randomly allocated into one of the three groups (7/each):

Group 1: zinc-carbonated nano-hydroxyapatite containing toothpaste (study group) Group 2: 8% arginine and calcium carbonate (Pro-Argin) containing toothpaste (study group) Group 3: fluoride containing toothpaste (positive control group)

Materials used in the study:

1. zinc-carbonated nano-hydroxyapatite containing toothpaste.
2. 8% arginine and calcium carbonate (Pro-Argin) containing toothpaste
3. fluoride containing toothpaste

   - Clinical procedures:

All interventions will be performed by the primary investigator as follows:

The dental plaque deposit will to be removed before the assessment. Dental prophylaxis will be performed with a bristle brush and non-fluoridated prophylactic paste during the initial clinical examination and before any examination.

photographic assessment by digital camera will be performed at 0 , 3 months, and 6 months throughout the study period for all the patients. During the photographic assessment, all the photographs will be taken under fixed conditions using a digital camera with lens equipped with external ring flash with 1:1 shooting power. the image quality will be set as RAW format, the shutter speed will set to 1/125 sec, F22 aperture value, auto white balance, and ISO 200. All images will be saved as Joint Photographic Experts Group (JPEG) files suitable for manipulation with the image analysis software.

At the baseline of the study, all participants will be provided with instructions to adhere to strict oral hygiene practices. These instructions included brushing their teeth twice a day using the allocated toothpaste and a soft-bristle toothbrush, employing the Bass Technique for a duration of 1 to 2 minutes.Participants will be instructed to spit out the excess toothpaste rather than rinse their mouths with water after brushing with toothpaste.

Patient's confidentiality will be respected through the photographic technique.

After digital images captured, they will be downloaded and stored as JPEG. Then the size of each WSL will be analyzed, and compared with baseline lesions by using Abode Photoshop and ImageJ analysis softwares.

The enamel color of each WSL will be measured using the Standardized CIE Lab* system (Commission International de l'Eclairage) within Adobe Photoshop software.

All measurements will be performed under standardized ambient conditions to ensure accuracy and reproducibility.

- Follow up

Patients will be recalled after 1, 3, and 6 months for clinical examinations and photographic assessments and oral hygiene instructions will be further provided.

- Outcome measurement:

Photographic assessment for size and color change reading outcomes will be assessed by one calibrated examiners at the following periods:

1) Baseline 2) 3-month evaluation 3) 6-month evaluation

Photographic assessment:

The following will be determined from photographs of all the patients in relation to WSLs:

* Size readings The area of the labial surface of the tooth WSL area The area of WSL to area of the labial surface of the tooth ratio percent (Percent of WSL) The percentage of decrease in WSL ratio due to time (Percent Decrease)
* Color change readings The values of L* (differences in lightness ranging from O (black) to 100 (white)), a* (green-red coordinate), and b* (blue yellow coordinate) will be recorded for the WSL and the adjacent sound enamel.

Color change will be calculated as the color difference between the treated and untreated enamel, as well as the color difference between the WSL at baseline and at the different follow-up intervals.

- Degree of WSL masking after the treatment will be measured.

14 image will be re-examined after 1 weeks for intra-examiner reliability

in-vitro part: experimental study where a total of 36 sound premolars will be randomly allocated according to the assigned toothpaste into four groups: G1: zinc-carbonated nano-hydroxyapatite; G2: arginine; G3: positive control (fluoride toothpaste); and G4: negative control (artificial saliva). A scanning electron microscope (SEM) and energy dispersive X-ray (EDX) analysis will be conducted at the baseline to assess the calcium (Ca) and phosphorus (P) content. Following the induction of white spot lesions, a pH cycle will be implemented, involving a 7-day application of the toothpastes. Readings will be taken both after demineralization and subsequent remineralization phases.

ELIGIBILITY:
Inclusion Criteria:

* Completion of fixed appliance therapy within the past 1 week.
* Presence of at least one post-orthodontic white spot lesion on the labial surfaces of the six maxillary anterior teeth with a score of 1 or 2 on International Caries Detection and Assessment System (ICDAS II).

Exclusion Criteria:

* Previous or planned treatment of WSLs.
* Cavitated enamel surface.
* Teeth with any composite restorations, veneers, crowns.
* Surface defects (developmental defects, fluorosis, intrinsic and extrinsic discolorations, etc.).
* Smoking habits.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
the size | 1) Baseline 2) 3-month evaluation 3) 6-month evaluation
  Photographic assessment of the images will be done for quantifying the size (in mm2) of the white spot lesions and the affected tooth's labial surface by using an image processing software, ImageJ analysis software and to ensure accuracy of values, image calibration will be carried out, and the scale of the image analysis software will be pre-set. After the software calculates the values of the entire area of the tooth and the size of the WSL, the area affected by white spot lesions will be expressed as a percentage of the total tooth surface: WSLs %= Area of WSL/ Area of the labial tooth surface*100.
the color change | 1) Baseline 2) 3-month evaluation 3) 6-month evaluation
  Using the Standardized CIE Lab* system within Adobe Photoshop software, L*a*b values will be analyzed for each tooth and the color changes between carious and healthy enamel (∆E*ab), as well as changes between different time points (∆E*ab), will be calculated by = Δ E = (Δ L 2 + Δ a2 + Δ b2) ½. ΔE values between 1 and 3.7 are not only acceptable but also often go unnoticed in various colors, especially darker shades. Conversely, when ΔE exceeds 3.7, the color change could be clinically visible, indicating a noticeable color mismatch. According to the degrees of color changes evaluated 6 months after treatment, the teeth will be divided into the following three types:
  Type 1: The whitish, opaque color is completely masked Type 2: The whitish opaque color is partially masked but not completely Type 3: The whitish opaque color shows little

SECONDARY OUTCOMES:
Evaluation of the remineralizing ability of each agent | 1 month
  assessing Calcium (Ca) and Phosphorus (P) in weight percentage and Ca/P ratio for all groups by using Energy dispersive X-ray Spectroscopy (EDX) Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schlagenhauf U, Kunzelmann KH, Hannig C, May TW, Hosl H, Gratza M, Viergutz G, Nazet M, Schamberger S, Proff P. Impact of a non-fluoridated microcrystalline hydroxyapatite dentifrice on enamel caries progression in highly caries-susceptible orthodontic patients: A randomized, controlled 6-month trial. J Investig Clin Dent. 2019 May;10(2):e12399. doi: 10.1111/jicd.12399. Epub 2019 Jan 30. PMID 30701704
- [Background] Butera A, Pascadopoli M, Gallo S, Lelli M, Tarterini F, Giglia F, Scribante A. SEM/EDS Evaluation of the Mineral Deposition on a Polymeric Composite Resin of a Toothpaste Containing Biomimetic Zn-Carbonate Hydroxyapatite (microRepair(R)) in Oral Environment: A Randomized Clinical Trial. Polymers (Basel). 2021 Aug 16;13(16):2740. doi: 10.3390/polym13162740. PMID 34451279